CLINICAL TRIAL: NCT02726802
Title: Effectiveness of Two Different Entry Portal Pathways Into Primary Care for Musculoskeletal Injury: A Randomized Controlled Trial
Brief Title: Effectiveness of Two Different Entry Portal Pathways Into Primary Care for Musculoskeletal Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Reynolds Army Community Hospital (U.S. Federal Agency)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); Temple University (Other)
Responsible Party: Principal Investigator, Kathryn M. O'Bright (Finn), DPT, OCS, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 413803-1
Record Dates: First submitted 2016-01-11; First posted 2016-04-04 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Physical Therapy Direct Access; Physical Therapy Primary Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Physical Therapy route of entry (Experimental): The subject will see a physical therapist as their initial encounter into the healthcare system
  Interventions: Other: physical therapy vs. primary care interventions
- Primary Care Provider rout of entry (Active Comparator): The subject will see a primary care provider as their initial encounter into the healthcare system
  Interventions: Other: physical therapy vs. primary care interventions

INTERVENTIONS:
Other: physical therapy vs. primary care interventions — Subjects with acute (< 3 months onset) will be randomized to see either a physical therapist or a primary care provider as their initial entry into the healthcare system

SUMMARY:
This study aims to compare the self-report functional outcome measures, medical readiness and healthcare utilization (overall cost of imaging, prescription medications for pain, and follow-up visits) of soldiers with musculoskeletal injuries first seen by a physical therapist versus primary care provider.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 18
* Musculoskeletal injury or complaint < 3 months since onset
* Active duty service member, reachable by phone/e-mail within 3 months of initial encounter

Exclusion Criteria:

* Subject currently has a permanent profile for any reason OR subject has a temporary profile for a body part in the same half of the body as the current complaint OR solider is pending physical examination board (PEB) or undergoing/pending medical examination board (MEB)
* Individuals undergoing PEB/MEB are made aware that the end-state of the process includes a certain percentage of government monetary compensation based on their physical or mental disability, i.e, higher disability equates to greater pay. Because of this, individuals may be motivated to demonstrate worse outcomes as it may result in a higher disability "rating". For this reason, these individuals will be excluded from the study.
* Subject has been treated previously for the same condition within the past 3 months
* Subject has history of surgery for the same body part within the past 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Patient Specific Functional Scale | 3 months
PROMIS physical function scale | 3 months
Global Rating of Change (GROC) | 3 months
Defense and Veterans Pain Rating Scale | 3 months

SECONDARY OUTCOMES:
Self-Report Medical Readiness Questionnaire | 3 months
  This questionnaire consists of 6 questions that ask the patient to rate their ability to perform various soldier/deployment-related tasks. This will provide way of measuring the soldier's perceived status of medical readiness before and after episodes of medical care.
Medical Profile Status | 3 months
  The medical profile is the Army's assessment of a soldier's overall medical readiness, i.e.: deployability. A profile for musculoskeletal injury can be temporary (T) or permanent (P) and deployable (2) or non-deployable (3). The profile is used to limit the soldier's activities to accommodate their injury or complaint. Evaluating the medical profile status in this study will serve as a way to measure the subjects' medical readiness.
Overall Healthcare Consumption | 12 months
  overall healthcare consumption as measured by the dollar-value of each medical encounter following the initial encounter
Patient Satisfaction | 3 months
  Likert Scale 0-10, how satisfied is the patient with the care they received.
Report of adverse events | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Reynolds Army Community Hospitral, Fort Sill, Oklahoma, United States